CLINICAL TRIAL: NCT02634216
Title: Effects of Capros Supplementation on Hyperglycemia in Patients With Type-1 Diabetes
Brief Title: Effects of Capros in Patients With Type-1 Diabetes
Acronym: CarposT1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Natreon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014H0206
Record Dates: First submitted 2015-06-26; First posted 2015-12-17 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Type I Diabetes
Keywords: Hyperglycemia; Capros; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type 1 Diabetics using CGM (Experimental): Type 1 diabetics using Continuous Glucose MonitoringCGM to take 500 mg daily of Capros supplement (250 mg twice a day) at lunch and dinner.
  Interventions: Dietary Supplement: Capros

INTERVENTIONS:
Dietary Supplement: Capros — 250 mg BID

SUMMARY:
The purpose of this 12 week longitudinal study is to test the effect of the dietary supplement, Capros, on blood glycemic index of Type 1 diabetics that have a sensor that provides continuous glucose monitoring (CGM). 20 Type 1 Diabetics will take the Capros supplement for 12 weeks to determine the effect of blood glycemic index. Capros, is a generally safe dietary supplement currently sold over the counter in the United States. Type 1 diabetes also known as juvenile diabetes is commonly diagnosed in children and young adults. Insulin is converted into energy needed for daily living, and with diabetes, insulin is not produced in the body as it should causing many problems. In traditional Indian medicine, the gooseberry Phyllanthus emblica has been used for thousands of years as an effective source of polyphenols and antioxidants. A 12 week longitudinal study to determine the effect of the dietary supplement, Capros, on the blood glycemic index in patients with Type 1 diabetes (T1D).

DETAILED DESCRIPTION:
There are a total of 4 study visits,over the course of 12 weeks. These visits will occur on weeks 1, 4, 8, and 12. At each study visit the the following will be recorded: Age, Sex, Pulse, height, weight, CGM real time measurement and the following non-medical information will be recorded: Address, Phone number and Email address ( will be recorded at the first visit and will be asked if anything has changed at the reoccurring visits). The following will happen at each visit:

Visit 1 (Week 0): The subject will be presented with informed consent. Data will be collected on a data collection sheet, a finger stick for A1C will be obtained (if not completed as SoC), Continuous Glucose Monitoring will be downloaded, UPT for WCBP will be performed, the subject will be given a 4-week supply of the Capros supplement and a subject diary. The subject will be given a subject diary to document their morning/evening sugar and the time of when participants take the supplements. The subject will be asked to bring in the diary to each follow-up visit to check for compliance verification.

Visit 2 and 3 (Week 4 and 8): The following activities will take place during these visits: AE review, concomitant medications review, weight, vital signs, CGM download, pill count and distribution, collect previous diary and provide new.

Visit 4 (Week 12): The following activities will take place during these visits: AE review, concomitant medications review, weight, vital signs, CGM download, pill count, collect previous diary. Also, at this visit, a finger stick for A1C (if not completed as SoC), no further distribution of supplements.

Taking the supplement: After receiving the supplement, the subject is instructed to take 2 capsules per day by mouth, once with food around lunchtime and once with food around dinner time for a total of 12 weeks. The subjects will be asked to keep all empty bottles/ any remaining Capros supplements and bring them to each follow-up visit for a compliance check. Participants will receive a new 4-week supply of supplements at study visits 2 and 3.

Risks for participating in this study are extremely low. Capros is a dietary supplement derived from the Indian Gooseberry, and contains no artificial ingredients, is non-toxic and is safely tolerated among humans. Capros is currently sold over the counter in the U.S. and has no known side effects; however an allergic reaction to the supplement is possible.

There is a potential risk for hypoglycemia while taking this supplement. In the even that this occurs, subjects are instructed to follow their primary care physician instructions for this and record it on their data log.

This is not a treatment study so subjects may have no direct benefit while taking the supplement. The investigators are looking to monitor and observe if any changes take place with participants blood sugar level over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 10 - 60 yrs. of age
* Type 1 Diabetes using Continuous Glucose Monitoring (CGM) for at least the last 3 months
* Less than 10% variation in prescribed long acting dosages in the previous 3 months

Exclusion Criteria:

* Individuals who are deemed unable to understand the procedures, risks and benefits of the study, i.e. informed consent will be excluded from the study
* Females who are pregnant
* Individuals who are therapeutically immuno-compromised
* Prisoners
* Anyone with a known allergy to amla fruit
* Current use of any of the following medications will result in exclusion:
* Steroids (Prednisone, etc.)
* Immunosuppressants
* Accutane (last 6 months)

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Effect of Capros on Blood Glycemic Index | 12 weeks
  To determine the effect on blood glycemic index in Type 1 Diabetics with taking the nutritional supplement Capros

CONTACTS AND LOCATIONS:
Overall Officials: Gayle M. Gordillo, M.D., Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Carepoint East 543 Taylor Ave., Columbus, Ohio
  - Martha Morehouse Medical Plaza 2050 Kenny Road, Columbus, Ohio
  - Davis Heart and Lung Research Institute, Columbus, Ohio

REFERENCES:
- [Result] Hiraganahalli BD, Chinampudur VC, Dethe S, Mundkinajeddu D, Pandre MK, Balachandran J, Agarwal A. Hepatoprotective and antioxidant activity of standardized herbal extracts. Pharmacogn Mag. 2012 Apr;8(30):116-23. doi: 10.4103/0973-1296.96553. PMID 22701284
- [Result] Sabu MC, Kuttan R. Anti-diabetic activity of medicinal plants and its relationship with their antioxidant property. J Ethnopharmacol. 2002 Jul;81(2):155-60. doi: 10.1016/s0378-8741(02)00034-x. PMID 12065146